CLINICAL TRIAL: NCT06103058
Title: The Prevalence of Fibromyalgia in Adults at Al-Karak Jordan a Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Mohammad Abu-Jeyyab, Mutah university, Mutah University
Other Study IDs: 20235012
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Fibromyalgia; Orthopedic Disorder
MeSH Terms: conditions — Fibromyalgia; Musculoskeletal Diseases | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for fibromyalgia: 26.5% prevalence of fibromyalgia
- Negative for fibromyalgia: 26.5% prevalence of fibromyalgia
  Interventions: Other: Cross sectional

INTERVENTIONS:
Other: Cross sectional — Cross sectional
  Groups: Negative for fibromyalgia

SUMMARY:
Fibromyalgia is a chronic and intricate musculoskeletal disorder characterized by widespread pain, fatigue, and tenderness in specific anatomical regions. Although its prevalence varies among populations, understanding the prevalence in different geographical areas is crucial for healthcare planning. This cross-sectional study aims to determine the prevalence of fibromyalgia in adults residing in Al-Karak, Jordan. The city's unique demographic and environmental characteristics may influence the occurrence of fibromyalgia among its adult population. The study aims to address gaps in knowledge, provide localized insights, and shed light on fibromyalgia's burden on the community's health. Accurate prevalence data aids healthcare planning and resource allocation.

ELIGIBILITY:
Using google forms, this cross-sectional study was carried out, and the participants were reached via social media platforms (5)

. Participants' autonomy was maintained, and no direct benefit was gained in return for filling out the questionnaire. The ethics committee at the Faculty of Medicine, Mutah University, Karak, Jordan, provided the required ethical approval prior to the initiation of this study. Moreover, the committee ensured that the study was designed according to the principles of the Declaration of Helsinki (Date: 13 February 2023. Reference number: 992023). In this study, the authors targeted Karak government citizens, in Jordan. Accordingly, the required sample size to achieve a 99% Confidence interval was 663 participants.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study found a 26.5% prevalence of fibromyalgia in the studied population. Female gender, mental health illnesses, and comorbidities like irritable bowel syndrome, psychiatric disorders, and rheumatological and neurological diseases were significantly associated with fibromyalgia. Age, BMI, marital status, employment status, and certain comorbidities did not show statistically significant predictive value.
  Discussion: The significant prevalence of fibromyalgia and its links to female gender, mental health problems, and comorbidities highlight the necessity for specific healthcare interventions and public awareness initiatives. The study's findings help to understand the imp
Sampling Method: Probability Sample
Enrollment: 965 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cross sectional | 2 years
  Outcome measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Mutah University, Qīr Moāv, Jordan

IPD SHARING:
Plan to Share IPD: Undecided